CLINICAL TRIAL: NCT02815787
Title: A Single Randomized, Open, Cross-over, Phase Ie Study to Access the Drug-drug Interaction of SP2086 and Glyburide
Brief Title: The Drug -Drug Interaction of SP2086 and Glyburide
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: QLHCPI-179
Record Dates: First submitted 2016-01-03; First posted 2016-06-28 (Estimated); Last update posted 2016-06-28 (Estimated); Status verified 2016-06

CONDITIONS: Type 2 Diabetes
Keywords: SP2086; Glyburide; drug-drug interaction
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Glyburide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SP2086 and Glyburide (Active Comparator): The A sequence was that Glyburide was taken at 5mg qd dose on Days1,4,5,6,7 and 8; SP2086 will be administered orally (by mouth) as 200mg on Days 8.The B sequence was that SP2086 was taken at 200mg qd dose on Days1,4,5,6,7 and 8;Glyburide will be administered orally (by mouth) as 200mg on Days 8.The trial period were 25 days. In this group,the subjects was given the drugs from A sequence to the B sequence.
  Interventions: Drug: SP2086; Drug: Glyburide
- Glyburide and SP2086 (Active Comparator): The A sequence was that Glyburide was taken at 5mg qd dose on Days1,4,5,6,7 and 8; SP2086 will be administered orally (by mouth) as 200mg on Days 8.The B sequence was that SP2086 was taken at 200mg qd dose on Days1,4,5,6,7 and 8;Glyburide will be administered orally (by mouth) as 200mg on Days 8.The trial period were 25 days.In this group,the subjects was given the drugs from B sequence to the A sequence.
  Interventions: Drug: SP2086; Drug: Glyburide

INTERVENTIONS:
Drug: SP2086 — In the A sequence Glyburide was taken at 5mg qd dose on Days1,4,5,6,7 and 8; SP2086 will be administered orally (by mouth) as 200mg on Days 8.In the B sequence was that SP2086 was taken at 200mg qd dose on Days1,4,5,6,7 and 8;Glyburide will be administered orally (by mouth) as 200mg on Days 8.
Drug: Glyburide — In the A sequence Glyburide was taken at 5mg qd dose on Days1,4,5,6,7 and 8; SP2086 will be administered orally (by mouth) as 200mg on Days 8.In the B sequence was that SP2086 was taken at 200mg qd dose on Days1,4,5,6,7 and 8;Glyburide will be administered orally (by mouth) as 200mg on Days 8.

SUMMARY:
The purpose of the study is to investigate the potential interaction between SP2086 and Glyburide after the singe and multiple oral doses treatment in healthy adult volunteers respectively.

DETAILED DESCRIPTION:
This is an open-label (volunteers will know the names of treatments they are assigned) single-center and cross-over study of SP2086 and Glyburide in healthy adult volunteers. All subject were randomized into two groups, and the drugs will be administered according to the AB and BA sequences.The A sequence was that Glyburide was taken at 5mg qd dose on Days1,4,5,6,7 and 8; SP2086 will be administered orally (by mouth) as 200mg on Days 8.The B sequence was that SP2086 was taken at 200mg qd dose on Days1,4,5,6,7 and 8; Glyburide will be administered orally (by mouth) as 200mg on Days 8.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers with a body mass index(BMI) between 19 and 24 Kg/m2
* Had signed the informed consent himself or herself.

Exclusion Criteria:

* Have the abnormal lab or other examination results and the change have clinical significance.
* Known allergy to SP2086 or Glyburide or any of the excipients of the formulation of SP2086 or Glyburide.
* History of using the sulfa or sulfonylureas or DPP-IVor GLP-1 drugs or other similar structure drugs.
* History of severe unconsciousness hypoglycemia
* History of any surgery prior to screening in 6 months.
* History of blood donation≥400 mL prior to screening in 3 months or participate in blood donation,or by blood transfusion in one month.
* History of participate any drug or medical device prior to screening in 3 months.
* Within a month before the screening using any prescription drugs, over-the-counter drugs, Chinese herbal medicine (especially oral antidiabetics drugs) or food supplements( vitamins).
* 2 days before the randomization ,the patients can not ban alcohol, tobacco, or reference food or drink containing caffeine or xanthine , or vigorous exercise, or there are other factors that can affect drug absorption, distribution, metabolism and excretion.
* The hepatitis B surface antigen, hepatitis c antibody, HIV antibody and syphilis antibody was positive.
* Pregnancy or lactation women, or a fertility male or female is not willing to contraception during test.
* Researchers considered that there was any situation that may cause the participants can't finish this study or bring any obvious risk to subjects.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2014-03; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
The maximum plasma concentration (Cmax) of SP2086 | up to Day 25
  Cmax (a measure of the body's exposure to SP2086) will be compared before and after administration of multiple doses of SP2086
The maximum plasma concentration (Cmax) of SP2086 acid | up to Day 25
  Cmax (a measure of the body's exposure to SP2086 acid) will be compared before and after administration of multiple doses of SP2086
The maximum plasma concentration (Cmax) of Glyburide | up to Day 25
  Cmax (a measure of the body's exposure to Glyburide) will be compared before and after administration of multiple doses of Glyburide
The area under the plasma concentration-time curve (AUC) of SP2086 | up to Day 25
  AUC (a measure of the body's exposure to SP2086) will be compared before and after administration of multiple doses of SP2086
The area under the plasma concentration-time curve (AUC) of SP2086 acid | up to Day 25
  AUC (a measure of the body's exposure to SP2086 acid) will be compared before and after administration of multiple doses of SP2086
The area under the plasma concentration-time curve (AUC) of Glyburide | up to Day 25
  AUC (a measure of the body's exposure to Glyburide) will be compared before and after administration of multiple doses of Glyburide

SECONDARY OUTCOMES:
The number of volunteers with adverse events as a measure of safety and tolerability | up to Day 25

CONTACTS AND LOCATIONS:
Overall Officials: RuiChen Guo, M.D, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China